CLINICAL TRIAL: NCT06351553
Title: Effect of the Autonomic Nervous System on the Outcomes of PULSEd Field Ablation to Treat Atrial Fibrillation (EASy-PULSE AF)
Brief Title: Effect of the Autonomic Nervous System on the Outcomes of PULSEd Field Ablation to Treat Atrial Fibrillation
Acronym: EASy-PULSE AF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Jose Luis Ibañez Criado, Principal Investigator, Hospital General Universitario de Alicante
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-169
Record Dates: First submitted 2024-03-13; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Pulmonary Vein Isolation; Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pulmonary vein isolation exclusively with radiofrequency (Active Comparator): The ablation of the anterior and posterior wall will be performed with radiofrequency.
  Interventions: Procedure: Pulmonary vein isolation exclusively with radiofrequency
- Pulmonary vein isolation exclusively with pulsed field ablation (Experimental): The ablation of the anterior and posterior wall will be performed with pulsed field ablation.
  Interventions: Procedure: Pulmonary vein isolation exclusively with pulsed field ablation
- Combined pulmonary vein isolation (Experimental): The ablation of the anterior wall will be performed with radiofrequency, and the posterior wall with pulsed field ablation.
  Interventions: Procedure: Combined pulmonary vein isolation

INTERVENTIONS:
Procedure: Pulmonary vein isolation exclusively with radiofrequency — The QDOT (Biosense Webster, Inc.) or TactiFlex (Abbott S.E.) catheters will be used. The ablation will be controlled by temperature, with a limit of 42ºC and a power target of 30-40W. A high-power strategy (90 W/4 seconds) can be used on the posterior wall when the QDOT catheter is used.
  Arms: Pulmonary vein isolation exclusively with radiofrequency
Procedure: Pulmonary vein isolation exclusively with pulsed field ablation — The Sphere-9 catheter will be used (with biphasic and unipolar wave), with a duration per application of 5 seconds and a separation between lesions of 5-6mm. The target temperature increase will be at least 1.5ºC above the patient's basal temperature to mark the ablation as effective.
  Arms: Pulmonary vein isolation exclusively with pulsed field ablation
Procedure: Combined pulmonary vein isolation — The Sphere-9 catheter will be used for both radiofrequency and pulsed field ablation. When using radiofrequency, the ablation will be temperature controlled, with a target temperature of 73ºC. The duration per application will be 5 seconds. Catheter irrigation during ablation will be 30ml/min, with a maximum current intensity of 3700mA, and a maximum current density of 13.6mA/mm2. The separation between lesions will be 7-8mm. Regarding pulsed field ablation, the characteristics will be those indicated in "Pulmonary vein isolation exclusively with pulsed field ablation" group.
  Arms: Combined pulmonary vein isolation

SUMMARY:
Pulmonary vein (PV) isolation is considered the therapeutic strategy of choice to maintain sinus rhythm (SR) in symptomatic patients with atrial fibrillation (AF). The most commonly used energy modality is radiofrequency (RF). However, this type of energy presents notable challenges, such as its lack of selectivity for myocardial tissue, which increases the risk of serious complications such as atrioesophageal fistula, PV stenosis, and vagus nerve injuries. In this context, PV isolation using pulsed field ablation (PFA) emerges as a promising alternative due to its greater myocardial selectivity. However, this selectivity presents additional challenges. Preliminary studies indicate that PFA may not damage the autonomic nervous system (ANS) involved in the initiation and maintenance of AF in certain patients, although stronger evidence is needed to support this claim.

The investigators propose to carry out a single-center clinical trial, although with the possibility in the future of including other centers. Patients will be randomized to three research groups: PV isolation with RF, PV isolation with PFA, and PV isolation combining PFA and RF (using RF on the anterior wall and PFA on the posterior wall). This assignment will be open to the operator who performs the procedure, but blind for the researcher responsible for monitoring and for the data analyst. The objective is to compare the impact of different energy sources during PV isolation on the ability to produce a permanent alteration in the ANS. The hypothesis is that combined PF isolation will be capable of producing a permanent alteration of autonomic function parameters superior to ablation using exclusive PFA.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a diagnosis of paroxysmal atrial fibrillation, referred to our center for pulmonary vein isolation, who are willing and able to sign the informed consent.

Exclusion Criteria:

* Patients with permanent atrial fibrillation.
* Patients with previous pulmonary vein isolation procedure.
* Patients with pacemakers, or with a diagnosis of atrioventricular block or sinus dysfunction.
* Patients who show their refusal to participate in the registry, or are unable to understand the informed consent.
* Patients under 18 years of age.
* Pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy primary outcome: Alteration of autonomic function parameters | Two years
  Determine if combined pulmonary vein isolation (anterior wall ablation with radiofrequency and posterior wall ablation with pulsed field ablation) will be capable of producing a permanent alteration of autonomic function parameters (average heart rate) greater than exclusive pulsed field ablation.

SECONDARY OUTCOMES:
Efficacy secondary outcome: Alteration of autonomic function parameters | Two years
  Determine if combined pulmonary vein isolation (anterior wall ablation with radiofrequency and posterior wall ablation with pulsed field ablation) will be capable of producing a permanent alteration of autonomic function parameters (attenuation of heart rate variability) greater than exclusive pulsed field ablation.
Efficacy secondary outcome: Alteration of autonomic function parameters | Two years
  Determine if combined pulmonary vein isolation (anterior wall ablation with radiofrequency and posterior wall ablation with pulsed field ablation) is at least as effective as exclusive radiofrequency pulmonary vein isolation in its ability to produce a permanent alteration of autonomic function parameters (average heart rate).
Efficacy secondary outcome: Alteration of autonomic function parameters | Two years
  Determine if combined pulmonary vein isolation (anterior wall ablation with radiofrequency and posterior wall ablation with pulsed field ablation) is at least as effective as exclusive radiofrequency pulmonary vein isolation in its ability to produce a permanent alteration of autonomic function parameters (attenuation of heart rate variability).
Efficacy secondary outcome: Procedure duration. | Two years
  Determine if combined pulmonary vein isolation or exclusive pulmonary vein isolation with pulsed field ablation will shorten procedure times compared to exclusive radiofrequency pulmonary vein isolation.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura García Cano, Alicante, Spain